CLINICAL TRIAL: NCT01410981
Title: Prognostic Potential of Cell Surface Markers and Pim Kinases in Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 101565
Record Dates: First submitted 2011-07-13; First posted 2011-08-05 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The patients will not have bone marrow biopsy or aspirate solely for this study. When the patients undergo routine bone marrow aspirate and biopsy for the purpose of initial diagnosis, followup or restaging, they will be asked and consented for participation in the study. The patient will then be treated with standard chemotherapy including Bortezomib-based, Revlimid-based, Thalidomide-based chemoregimen. The bone marrow aspirate from patients who consent to be in the study will be stained for CXCR4, CD47, pS6, in addition to standard study flow cytometry panel for multiple myeloma. The staining and flow cytometry analysis will be performed at the Clinical Flow Cytometry Facility (Director: Dr. Sally Self) according to the standard flow cytometry procedure. Sphingolipid gene expression levels will be measured. A small aliquot may be sent to collaborators in Genentech Corp for measurement of pS6 and Pim kinase expression. The sample information will be de-identified.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Multiple Myeloma subjects with bone marrow aspirate/biopsy: All patients seen at MUSC with a diagnosis of multiple myeloma or possible multiple myeloma who undergo bone marrow aspirate and biopsy will be approached for participation in this study.

SUMMARY:
The purpose of this study is to understand if small proteins found on the surface of myeloma cells (called CXCR4 and CD47) or inside the myeloma cells (Pim kinases, sphingolipids, and pS6) can predict how patients will respond to chemotherapy-treatment and if a small molecule inside the myeloma cells (called Pim kinase) can be used as a treatment target for myeloma. A sample from the bone marrow biopsy (a small amount of tissue removed from the body for laboratory testing) and aspirate (a small amount of fluid is removed from the body for laboratory testing) that had been done before the subject entered this study will be provided for research purposes. Based on preliminary data, it is hypothesized that CXCR4, CD47, sphingolipids, and Pim kinases could be used as prognostic/predictive markers and that Pim kinase inhibitors provide a new agent for the treatment of multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of multiple myeloma or possible multiple myeloma who will have a bone marrow biopsy and aspirate
* Planned therapy with standard chemotreatment for multiple myeloma
* Laboratory data such as calcium, beta 2-microglobulin, albumin, creatinine and bone survey available for staging purpose.
* ≥18 years old

Exclusion Criteria:

* < 18 years old
* Patients who will not receive chemotreatment
* Patients whose treatment records are not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be three different population of patients: 1) newly diagnosed, 2) relapsed, 3) refractory multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Measure the expression levels of CXCR4, CD47, and pS6 by flow cytometry in myeloma patient's marrow aspirate | 3 years
  Our Aim 1 is to perform a corrective study to measure the expression levels of CXCR4, CD47, and pS6 by flow cytometry in myeloma patient's marrow aspirate and correlate their expression level with patients' treatment responses

SECONDARY OUTCOMES:
Determine if Pim kinase inhibitors or sphingosine kinase 2 inhibitors will inhibit patients' myeloma cells | 3 years
  Our aim 2 involves only in vitro cell culture system and in vivo animal models. We will measure the efficacy of Pim kinase inhibitors in inhibiting patients' myeloma cell growth in vitro using cell culture system. We will also determine the efficacy of Pim kinase inhibitors and sphingosine kinase 2 inhibitors in inhibiting tumor growth of patients' myeloma cells in animal models. We will measure the tumor size in animal models. Our Aim 2 does not involve any measurement of human myeloma patients. Therefore, measures of safety, tolerability etc in patients are not applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Sundaramoorthy P, Gasparetto C, Kang Y. The combination of a sphingosine kinase 2 inhibitor (ABC294640) and a Bcl-2 inhibitor (ABT-199) displays synergistic anti-myeloma effects in myeloma cells without a t(11;14) translocation. Cancer Med. 2018 Jul;7(7):3257-3268. doi: 10.1002/cam4.1543. Epub 2018 May 15. PMID 29761903
- [Derived] Venkata JK, An N, Stuart R, Costa LJ, Cai H, Coker W, Song JH, Gibbs K, Matson T, Garrett-Mayer E, Wan Z, Ogretmen B, Smith C, Kang Y. Inhibition of sphingosine kinase 2 downregulates the expression of c-Myc and Mcl-1 and induces apoptosis in multiple myeloma. Blood. 2014 Sep 18;124(12):1915-25. doi: 10.1182/blood-2014-03-559385. PMID 25122609